CLINICAL TRIAL: NCT06312813
Title: Pilot Studies Evaluating Use of Topical Imipramine and Amitriptyline in Reducing Ultraviolet B Light-Induced Redness in Patients With Rosacea
Brief Title: Evaluating Use of Topical Imipramine and Amitriptyline in Reducing Ultraviolet B Light-Induced Redness in Patients With Rosacea
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Wright State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2023-296
Record Dates: First submitted 2024-03-08; First posted 2024-03-15 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Rosacea
MeSH Terms: conditions — Rosacea | interventions — Imipramine; Amitriptyline

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Imipramine and Vehicle (Experimental): 4% imipramine and vehicle are applied on a 2x2cm2 area of the subject's cheek. The imipramine is applied on one side of the subject's face (cheek) and vehicle is applied on the other side.
  Interventions: Drug: Imipramine; Drug: Vehicle
- Amitriptyline and Vehicle (Experimental): 4% amitriptyline and vehicle are applied on a 2x2cm2 area of the subject's cheek. The amitriptyline is applied on side of the subject's face (cheek) and vehicle is applied on the other side.
  Interventions: Drug: Amitriptyline; Drug: Vehicle

INTERVENTIONS:
Drug: Imipramine — 4% imipramine
  Arms: Imipramine and Vehicle
Drug: Amitriptyline — 4% amitriptyline
  Arms: Amitriptyline and Vehicle
Drug: Vehicle — 0.1ml propylene glycol

SUMMARY:
Rosacea is a common skin condition associated with easy blushing and red face; many patients with rosacea react to sunlight with increased redness. The purpose of this study is to determine if the use of a topical medication will help reduce sunlight induced redness and irritation in patients with rosacea.

ELIGIBILITY:
Inclusion Criteria:

* Fitzpatrick Skin Type I - IIII
* Self-identified rosacea or no history of flushing/blushing for controls
* Able to provide medical history and list of medications -- control subjects will not be allowed to take medications that are known to be photosensitizers.

Exclusion Criteria:

* Using imipramine, amitriptyline or any other tricyclic antidepressant (oral or topical)
* Using topical anti-inflammatory (within 1 week) or systemic agents (e.g. prednisone)
* Large tattoos in the designated testing areas
* Tanning bed use within last 3 months
* Photodynamic Therapy or UCB treatments in past 3 months
* Female Subjects: pregnant or nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-02-27 (Actual); Primary Completion 2028-12-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Difference in redness of Ultraviolet B induced erythema with 4% imipramine | 10 minutes post-treatment
  Erythema change from baseline with 4% imipramine application in response to a low level of UVB are measured by using a mexameter device and thermal photography.
Difference in redness of Ultraviolet B induced erythema with 4% imipramine | 60 minutes post-treatment
  Erythema change from baseline with 4% imipramine application in response to a low level of UVB are measured by using a mexameter device and thermal photography.
Difference in redness of Ultraviolet B induced erythema with 4% imipramine | 120 minutes post-treatment
  Erythema change from baseline with 4% imipramine application in response to a low level of UVB are measured by using a mexameter device and thermal photography.
Difference in redness of Ultraviolet B induced erythema with 4% imipramine | 24 hours post-treatment
  Erythema change from baseline with 4% imipramine application in response to a low level of UVB are measured by using a mexameter device and thermal photography.
Difference in redness of Ultraviolet B induced erythema with 4% amitriptyline | 10 minutes post-treatment
  Erythema change from baseline with 4% amitriptyline application in response to a low level of UVB are measured by using a mexameter device and thermal photography.
Difference in redness of Ultraviolet B induced erythema with 4% amitriptyline | 60 minutes post-treatment
  Erythema change from baseline with 4% amitriptyline application in response to a low level of UVB are measured by using a mexameter device and thermal photography.
Difference in redness of Ultraviolet B induced erythema with 4% amitriptyline | 120 minutes post-treatment
  Erythema change from baseline with 4% amitriptyline application in response to a low level of UVB are measured by using a mexameter device and thermal photography.
Difference in redness of Ultraviolet B induced erythema with 4% amitriptyline | 24 hours post-treatment
  Erythema change from baseline with 4% amitriptyline application in response to a low level of UVB are measured by using a mexameter device and thermal photography.

SECONDARY OUTCOMES:
Tolerability of 4% imipramine on facial skin | 10 minutes post-treatment
  The tolerability of 4% imipramine on facial skin at baseline/Day 1 compared to Day 2 is measured by the Visual Analog Scale for pain and itch. [0= no skin pain/itch; 10 = severe skin pain/itch]
Tolerability of 4% imipramine on facial skin | 60 minutes post-treatment
  The tolerability of 4% imipramine on facial skin at baseline/Day 1 compared to Day 2 is measured by the Visual Analog Scale for pain and itch. [0= no skin pain/itch; 10 = severe skin pain/itch]
Tolerability of 4% imipramine on facial skin | 120 minutes post-treatment
  The tolerability of 4% imipramine on facial skin at baseline/Day 1 compared to Day 2 is measured by the Visual Analog Scale for pain and itch. [0= no skin pain/itch; 10 = severe skin pain/itch]
Tolerability of 4% imipramine on facial skin | 24 hours post-treatment
  The tolerability of 4% imipramine on facial skin at baseline/Day 1 compared to Day 2 is measured by the Visual Analog Scale for pain and itch. [0= no skin pain/itch; 10 = severe skin pain/itch]
Tolerability of 4% amitriptyline on facial skin | 10 minutes post-treatment
  The tolerability of 4% amitriptyline on facial skin at baseline/Day 1 compared to Day 2 is measured by the Visual Analog Scale for pain and itch. [0= no skin pain/itch; 10 = severe skin pain/itch]
Tolerability of 4% amitriptyline on facial skin | 60 minutes post-treatment
  The tolerability of 4% amitriptyline on facial skin at baseline/Day 1 compared to Day 2 is measured by the Visual Analog Scale for pain and itch. [0= no skin pain/itch; 10 = severe skin pain/itch]
Tolerability of 4% amitriptyline on facial skin | 120 minutes post-treatment
  The tolerability of 4% amitriptyline on facial skin at baseline/Day 1 compared to Day 2 is measured by the Visual Analog Scale for pain and itch. [0= no skin pain/itch; 10 = severe skin pain/itch]
Tolerability of 4% amitriptyline on facial skin | 24 hours post-treatment
  The tolerability of 4% amitriptyline on facial skin at baseline/Day 1 compared to Day 2 is measured by the Visual Analog Scale for pain and itch. [0= no skin pain/itch; 10 = severe skin pain/itch]

CONTACTS AND LOCATIONS:
Locations (1):
- Wright State Physicians, Fairborn, Ohio, United States